CLINICAL TRIAL: NCT02481856
Title: A Dose-response Evaluation of the SQ Tree SLIT-tablet in Subjects With Moderate to Severe Allergic Rhinoconjunctivitis Induced by Pollens From the Birch Group During Controlled Exposure in an Environmental Exposure Chamber
Brief Title: A Dose-response Evaluation of the SQ Tree SLIT-tablet Using an Environmental Exposure Chamber
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Collaborators: Inflamax Research Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TT-03
Record Dates: First submitted 2015-04-30; First posted 2015-06-25 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Allergic Rhinoconjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 12 DU SQ tree SLIT-tablet (Experimental): Betula verrucosa, allergen extract, Oral lyophilisate
  Interventions: Drug: SQ tree SLIT-tablet
- 7 DU SQ tree SLIT-tablet (Experimental): Betula verrucosa, allergen extract, Oral lyophilisate
  Interventions: Drug: SQ tree SLIT-tablet
- 2 DU SQ tree SLIT-tablet (Experimental): Betula verrucosa, allergen extract, Oral lyophilisate
  Interventions: Drug: SQ tree SLIT-tablet
- Placebo (Placebo Comparator): No active ingredient, Oral lyophilisate
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SQ tree SLIT-tablet
  Arms: 12 DU SQ tree SLIT-tablet; 2 DU SQ tree SLIT-tablet; 7 DU SQ tree SLIT-tablet
Drug: Placebo
  Arms: Placebo

SUMMARY:
The trial is a phase II, randomised, parallel-group, double-blind, placebo-controlled multi-site trial conducted in Canada. Before the start of treatment, the subjects will undergo baseline birch and oak Environmental Exposure Chamber sessions. The treatment duration is 24 weeks. The subjects will undergo birch Environmental Exposure Chamber sessions after 8, 16 and 24 weeks of treatment and an oak Environmental Exposure Chamber session after 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before any trial related procedures are performed
* Male or female aged 18 to 65 years
* Female subjects of child-bearing potential must have a negative urine pregnancy test and be willing to practise contraceptive methods
* History of moderate-to-severe rhinoconjunctivitis induced by pollens from the birch group with or without asthma despite having received treatment with symptom relieving medication during the previous 2 tree pollen seasons
* Positive SPT response (wheal diameter ≥ 3 mm) to Betula verrucosa
* Positive specific IgE against Bet v1 (≥ IgE Class 2; ≥0.70 kU/L)
* Willing and able to comply with the trial protocol
* Minimum level of rhinoconjunctivitis symptoms, defined as a TSS of at least 7 (of 18), at one timepoint during birch baseline EEC session.

Exclusion Criteria:

* Symptoms induced by interfering allergens that are expected to be present during the periods where the subject attends the EEC sessions
* Rhinoconjunctivitis caused by animal hair and dander to which the subject is regularly exposed.
* Allergic symptoms induced by perennial allergens such as house dust mites, and moulds
* A clinical history of uncontrolled asthma within 3 months prior to screening
* Reduced lung function FEV1 (< 70% of predicted value after adequate pharmacological treatment)
* Asthma requiring treatment with inhaled corticosteroid within the past 3 months prior to screening
* Previous treatment with any allergy immunotherapy product with tree pollen allergens or a cross-reacting allergen within the past 5 years
* Ongoing treatment with any allergy immunotherapy product
* Immunosuppressive treatment within 3 months prior to the screening visit
* Treatment with tricyclic antidepressants, catecholamine-O-methyltransferase inhibitors, mono amine oxidase inhibitors and beta-blockers
* Treatment with antidepressant medication with antihistaminic effect
* Treatment with antipsychotic medications with antihistaminic effect
* Treatment with anti-IgE drugs within 130 days/5 half-lives of the drug (which ever longest)
* Treatment with an investigational drug within 30 days/5 half-lives of the drug (which ever longest) prior to screening
* Severe oral inflammation or oral wounds at randomisation
* Symptoms of or treatment for upper respiratory tract infection, acute sinusitis, acute otitis media or other relevant infections that have not resolved 1-week prior to the baseline birch and oak Environmental Exposure Chamber sessions and at the randomisation visit
* Clinically relevant nasal polyps
* A history of paranasal sinus surgery
* A history of surgery of nasal turbinates
* A history of anaphylaxis with cardiorespiratory symptoms
* A history of recurrent (defined as two or more episodes) generalised urticaria during the last 2 years
* A history of drug-induced (incl. Allergy Immunotherapy) facial angioedema or a family (parents and siblings) history of hereditary angioedema
* Any clinically relevant chronic disease (≥3 months duration) that in the opinion of the investigator would interfere with the trial assessments or the safety of the subject
* An uncontrolled systemic disease affecting the immune system (e.g. insulin-dependent diabetes, autoimmune disease, immune complex disease, or immune deficiency disease whether acquired or not)
* A history of allergy, hypersensitivity or intolerance to the investigational medicinal product (except Betula verrucosa) or any of the symptomatic medications provided in this trial
* Being immediate family of the investigator or trial staff, defined as the investigator's/staff's spouse, parent, child, grandparent or grandchild.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Average total rhinoconjunctivitis symptom score | After 24 weeks of treatment
  The total rhinoconjunctivitis symptom score will measured during a birch pollen challenge in the Inflamax Environmental Exposure Chamber

SECONDARY OUTCOMES:
Average total rhinoconjunctivitis symptom score | After 8 and 16 weeks of treatment
  The total rhinoconjunctivitis symptom score will measured during a birch pollen challenge in the Inflamax Environmental Exposure Chamber
Average total rhinoconjunctivitis symptom score | After 24 weeks of treatment
  The total rhinoconjunctivitis symptom score will measured during an oak pollen challenge in the Inflamax Environmental Exposure Chamber
Adverse events | During the 24-weeks treatment period
  Adverse events will be grouped by number of treatment-emergent AEs and IMP-related AEs and will further summarised by treatment group and MedDRA SOC, MedDRA PT and broken down by severity, seriousness, action taken, time from first intake to AE and re-occurence after IMP administration
Vital signs | During the 24-weeks treatment period
Lung function measures | During the 24-weeks treatment period
  Forced expiratory volume in 1 second and peak flow measurements will be performed.
Changes in significant clinical safety laboratory values | Before and after the 24-weeks treatment period
  Standard haematology, biochemistry, urinalysis analysis will be performed for each subject before and after the 24-weeks treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Couroux, MD, Principal Investigator — Inflamax Research Incorporated
Locations (1):
- Inflamax Research Inc., Mississauga, Ontario, Canada

REFERENCES:
- [Derived] Biedermann T, Couroux P, Greve TM, Makela M. Safety of the standardized quality tree sublingual immunotherapy tablet: Pooled safety analysis of clinical trials. Allergy. 2021 Dec;76(12):3733-3742. doi: 10.1111/all.14882. Epub 2021 May 15. PMID 33905129